CLINICAL TRIAL: NCT06475573
Title: Effect of Fermented Dietary Fiber and Probiotics on the Intervention of Overweight/Obese Patients With Impaired Glucose Regulation
Brief Title: Fermented Dietary Fiber and Probiotics on Overweight/Obese Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2022-0946
Record Dates: First submitted 2024-06-21; First posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Impaired Glucose Regulation; Overweight and Obesity
Keywords: impaired fasting glucose; impaired glucose tolerance; overweight and obesity; dietary fiber; Probiotic
MeSH Terms: conditions — Overweight; Obesity; Glucose Intolerance

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Consume two 35g sachets of fermented dietary fiber probiotic solid beverages daily, replacing part of the staple food for lunch and dinner.
  Interventions: Dietary Supplement: dietary fiber probiotic beverages
- Control Group (Active Comparator): Consume two 35g sachets of convenient whole grain porridge daily, replacing part of the staple food for lunch and dinner.
  Interventions: Other: whole grain porridge

INTERVENTIONS:
Dietary Supplement: dietary fiber probiotic beverages — The intervention period lasted for 8 weeks. During this time, Participants received dietary guidance from researchers. The target energy intake was based on the limited energy diet model recommended in the "Chinese Guidelines for Medical Nutrition Therapy of Overweight/Obesity (2021)". Carbohydrates were to account for 55%-60% and fat for 25%-30% of total daily energy intake. Participants in experimental group consumed two 35g sachets of fermented dietary fiber probiotic solid beverages daily, replacing part of the staple food for lunch and dinner.
  Arms: Experimental group
Other: whole grain porridge — The intervention period lasted for 8 weeks. During this time, Participants received dietary guidance from researchers. The target energy intake was based on the limited energy diet model recommended in the "Chinese Guidelines for Medical Nutrition Therapy of Overweight/Obesity (2021)".Participants in control group consumed two 35g sachets of convenient whole grain porridge daily, replacing part of the staple food for lunch and dinner.
  Arms: Control Group

SUMMARY:
This study aims to investigate the efficacy of fermented dietary fiber and probiotics in improving glycemic control and associated metabolic parameters in overweight/obese IGR patients. The ultimate goal is to establish a clinically applicable nutrition intervention strategy for glucose tolerance impaired individuals.

DETAILED DESCRIPTION:
Impaired glucose regulation (IGR), encompassing impaired fasting glucose (IFG) and/or impaired glucose tolerance (IGT), represents a crucial stage in the progression to type 2 diabetes. Characterized by a state of compensatory glucose dysmetabolism, IGR is closely linked to overweight/obesity and can be reversed through lifestyle interventions. Timely intervention during this stage can promote weight loss, delay or prevent the onset and development of diabetes, and reduce the risk of cardiovascular diseases, chronic kidney disease, and all-cause mortality.

Current treatment approaches for overweight/obese IGR patients include dietary and physical activity modifications, pharmacotherapy, and bariatric surgery. However, individual responses to these interventions vary considerably. Dietary fiber, essential for maintaining normal gastrointestinal function, has been associated with an increased risk of various diseases, including colorectal cancer, cardiovascular diseases, obesity, metabolic syndrome, and type 2 diabetes, when consumed in inadequate amounts. Conversely, the gut microbiota plays a pivotal role in diabetes development and progression. Probiotics, potentially through the stimulation of short-chain fatty acid production and the induction of gut hormone secretion that influences blood glucose levels, may exert beneficial effects by enhancing immune modulation, increasing anti-inflammatory cytokine production, reducing intestinal permeability, and mitigating oxidative stress.

Therefore, this study aims to investigate the efficacy of fermented dietary fiber and probiotics in improving glycemic control and associated metabolic parameters in overweight/obese IGR patients. The ultimate goal is to establish a clinically applicable nutrition intervention strategy for glucose tolerance impaired individuals.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years old
* Meet the criteria for impaired glucose regulation according to the "Guidelines for the Prevention and Treatment of Type 2 Diabetes in China (2020 Edition)":

IFG: Fasting blood glucose ≥ 6.1 mmol/L and < 7.0 mmol/L IGT: 2-hour postprandial glucose ≥ 7.8 mmol/L and < 11.1 mmol/L

* Meet the Asia-Pacific criteria for overweight and obesity: 23 kg/m2 ≤ BMI
* Signed informed consent

Exclusion Criteria:

* Patients diagnosed with diabetes or currently undergoing diabetes treatment
* Patients who have received weight loss medication or surgery in the past 3 months
* Patients who are taking corticosteroids or thyroid hormones
* Patients with secondary obesity caused by endocrine, genetic, metabolic, or central nervous system diseases
* Patients with severe liver function or abnormal kidney function
* Patients with diseases that affect food digestion and absorption
* Patients with cardiovascular diseases, grade 3 hypertension, chronic hepatitis, malignant tumors, anemia, mental illness and memory disorders, epilepsy, etc.
* Patients with active tuberculosis, AIDS, and other infectious diseases
* Pregnant or breastfeeding women
* Patients with limb disabilities or other conditions that the clinical investigator deems inappropriate for participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
fasting blood glucose | Baseline and after 8-week intervention
  fasting blood glucose after an overnight fast
2-hour postprandial blood glucose | Baseline and after 8-week intervention
  2-hour postprandial blood glucose after 75g Glucose Tolerance Test

SECONDARY OUTCOMES:
Body weight | Baseline; after 4-week intervention; after 8-week intervention
  Body weight
body composition | Baseline; after 4-week intervention; after 8-week intervention
  body composition measured by Bioelectrical impedance analysis, including body fat percentage, visceral fat area, skeletal muscle mass
Lipid profile | Baseline and after 8-week intervention
  Total cholesterol, triglycerides, HDL, LDL

CONTACTS AND LOCATIONS:
Overall Officials: Pianhong Zhang, MD, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- The Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China